CLINICAL TRIAL: NCT01279226
Title: Radiofrequency Magnetic Induction Device for Use in Dermatologic Procedures for the Non-Invasive Treatment of Wrinkles and Rhytides
Brief Title: Investigation of Radiofrequency Device for Treatment of Wrinkles and Rhytides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rocky Mountain Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0310-0002A
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-10

CONDITIONS: Laxity of Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Auralevée device — Single treatment with Auralevée device.

SUMMARY:
The purpose of this pilot research study is to collect information on the safety and effectiveness of an experimental device intended to be used to improve the appearance of the skin by reducing the visibility of wrinkles and by reducing the looseness of skin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 21 years old,
* Apparently healthy,
* Informed consent signed by the subject.

Exclusion Criteria:

* Tobacco smokers,
* History of skin hypersensitivity,
* Current skin disorder or infection (e.g., herpes simplex),
* Prior cosmetic treatments to the face (e.g. Botox) or facial fillers (e.g. Restylane),
* Subjects with a pacemakers, internal defibrillators or electronically, magnetically, and mechanically activated implants,
* Subjects with implanted medical prostheses (such as clips, pins or plates) proximal to the treatment site,
* The current or recent use (within the past 12 months) of isotretinoin,
* Pregnancy or breast feeding,
* Insulin dependent diabetic subjects,
* Oxygen dependent subjects,
* Subjects with severe chronic illness, scleroderma, or lupus,
* Subjects with open sores or scars in the treatment region, or
* Subjects with ischemia in the treatment region.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Improved cosmesis | 2-6 timepoints from 4 days to 6 months
  Photographs of subjects before and after treatment will be scored and compared. Histology of skin samples may be used to assess deleterious events and elucidate the operative mechanism.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cooperrider, MD, Principal Investigator — Laser Treatment Center; Stephen Flock, PhD, Study Director — Rocky Mountain Biosystems, Inc.
Locations (1):
- Laser Treatment Center, Kirkland, Washington, United States